CLINICAL TRIAL: NCT01158209
Title: An Observational, Epidemiological Study on the Prevalence of Human Papillomavirus (HPV) Types in Women >= 18 Years of Age, in Egypt
Brief Title: An Observational, Epidemiological Study on the Prevalence of Human Papillomavirus Types in Women in Egypt
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113367
Record Dates: First submitted 2010-06-11; First posted 2010-07-08 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2011-10

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endocervical samples

GROUPS / COHORTS (1):
- Assessed cohort: Subjects attending out-patient health services for gynaecological examination.
  Interventions: Procedure: Endocervical samples

INTERVENTIONS:
Procedure: Endocervical samples — Endocervical samples collection during routine gynaecological examinations.

SUMMARY:
The purpose of the study is to determine the Human Papillomavirus (HPV) prevalence and HPV type distribution among women aged >= 18 years, attending out-patient health services for gynaecological examination and who agree to HPV testing in Egypt .

ELIGIBILITY:
Inclusion Criteria:

* Women >= 18 years of age attending a clinic for gynaecological examination.
* Women who agree to provide a cervical sample for human papillomavirus testing.
* Written informed consent obtained from the subject.

Exclusion Criteria:

* Referral for abnormal cervical sample at the current visit.
* Abundant menstrual bleeding or vaginal discharge not allowing appropriate screening to be performed.
* History of hysterectomy.
* Known diagnosis of immunosuppression, or patient on immunosuppressives.
* Pregnant women.
* Having received one or more doses of HPV vaccine prior to participating in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women >= 18 attending out-patient departments of primary, secondary or tertiary care centres for gynaecological examination and agreeing to provide a cervical sample for human papillomavirus testing.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of Human papillomavirus (HPV) DNA and of any of the HPV types among women undergoing cervical sample testing. | Average timeframe: 12 months

SECONDARY OUTCOMES:
Occurrence of HPV DNA and of any of the HPV types among women of different age-strata undergoing cervical sample testing | Average timeframe: 12 months
Behavioural risk factors assessed by behavioral questionnaire | At the single study visit (Day 0)
Assessing the awareness of HPV in relation to transmission and cause of cervical cancer | At the single study visit (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Egypt (2):
  - GSK Investigational Site, Alexandria
  - GSK Investigational Site, Cairo

REFERENCES:
- [Derived] Shaltout MF, Sallam HN, AbouSeeda M, Moiety F, Hemeda H, Ibrahim A, Sherbini ME, Rady H, Gopala K, DeAntonio R. Prevalence and type distribution of human papillomavirus among women older than 18 years in Egypt: a multicenter, observational study. Int J Infect Dis. 2014 Dec;29:226-31. doi: 10.1016/j.ijid.2014.07.029. Epub 2014 Nov 1. PMID 25447728